CLINICAL TRIAL: NCT00063843
Title: A Phase I, Dose-Escalating Study to Assess the Safety, Tolerability, and Immunogenicity of Recombinant Anthrax Protective Antigen Vaccine (rPA) Administered in Two Intramuscular Doses to Healthy Adults
Brief Title: Anthrax-rPA: Safety, Tolerability, Immunogenicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 01-003; Anthrax CVD 1000
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-05

CONDITIONS: Anthrax
Keywords: Bacillus anthracis (anthrax)
MeSH Terms: conditions — Anthrax | interventions — Anthrax Vaccines

INTERVENTIONS:
Biological: Recombinant Protective Antigen, Anthrax Vaccine Adsorbed

SUMMARY:
The primary objective is to determine the tolerability and safety, from days 0 to 210, of escalating doses of rPA either with or without Alhydrogel (an adjuvant; used to increase the action of the principle drug) given in a two-dose, intramuscular regimen to health adults. The secondary objective is to evaluate antibody responses to rPA, from days 0 to 210, following one of four escalating doses of vaccine given with and without Alhydrogel given in a two-dose series to healthy adults, and to compare immune responses following rPA with those following BioThrax (tm) given by either the intramuscular or SQ route. The tertiary objective is to describe the antibody kinetics following vaccination. This information will be used to determine the most probable optimal dose of rPA and/or Alhydrogel that is safe, well tolerated, and maximally immunogenic for use in future phase II trials.

DETAILED DESCRIPTION:
This Phase I, Dose-Escalating clinical study is designed to examine the immunologic response to rPA in the presence and absence of Alhydrogel at the 2 lowest dose levels. The study will investigate whether use of an aluminum-based adjuvant results in an increase in the magnitude or the duration of the antibody response, thus providing information on the necessity of aluminum-based adjuvants in formulations used in the phase II clinical trials. The rationale for the use of BioThrax by two administration routes in this trial is to allow for preliminary comparisons of the immune response following the currently available vaccine to the response following the new recombinant product. Approximately 80 outpatient community volunteers from the Baltimore-Washington area aged 18-40 years will be recruited on the basis of good health, expressed interest in the study, and availability for follow-up as determined at a preliminary interview. Each eligible subject will be enrolled in 1 of 4 study groups, each with three arms, for 7 months. The subjects' randomly assigned and double-masked to Arms A and B will have a 30 day screening period in which they will receive two doses of IM rPA or IM rPA+Alhydrogel or IM BioThrax one month apart, with follow up days on 1, 2, 7, 14, 28, 29, 30, 35, 42, 120, and 210. The subjects randomly assigned, but unmasked, to arms 1-C or 2-C will receive 3 doses of SQ BioThrax at 14 day intervals with follow up on days 1, 2, 7, 14, 15, 16, 21, 28, 29, 30, 35, 42, 120 and 210. The information gathered from the study objectives will be used to determine the most probable optimal doses of rPA +/- Alhydrogel that are safe, well tolerated, and maximally immunogenic for use in future phase II trials.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 40 years, inclusive. Good health as evidenced by screening evaluation within the 30 days prior to immunization. Expressed interest and availability to fulfill the study requirements. Signed, informed consents: screening, HIV antibody testing, stored specimen, HIPAA authorization, and protocol-specific consents. Agreement to avoid pregnancy for the 30 days following each vaccination by use of highly effective birth control methods. A highly effective birth control method is defined as one which results in a failure rate less than 1% per year when used consistently and correctly. These methods include tubal ligation, implants, injectables, combined oral contraceptives, some IUD's (All commonly used copper and hormone implanted IUD's in the US are highly effective including the following types: TCu-380A, TCu-220C, MLCu-375, Nova-T, and LNG-20. The less effective IUD's include the Lippes loop and the stainless steel ring), sexual abstinence, and a vasectomized partner. Agreement to refrain from taking any experimental drug or vaccine from day -30 to day 90.

Exclusion Criteria:

History of any of the following medical illnesses: Diabetes mellitus, Cancer, Heart disease (including hospitalization for heart attack, arrhythmia, or syncope), Unconsciousness (other than a single brief concussion), Seizures (other than simple benign febrile seizures of childhood), Gastrointestinal disease (including inflammatory bowel disease, celiac disease, and ulcers), Recurrent arthritis, Immunodeficiency, Autoimmune disease (including Systemic Lupus Erythematosus), Any current illness requiring daily medication (other than vitamins, contraceptives, and topical medications), Other conditions that in the opinion of the investigator would jeopardize the safety of the subject or the evaluation of the study objectives. Abnormal physical findings including, but not limited to, the following: Cardiac murmur (other than a functional murmur), Focal neurologic deficit, Hepatomegaly or splenomegaly, Lymphadenopathy, Jaundice, Hypertension (BP>150/90 on 2 separate days), Body mass index above 35 or below 19. Body mass index, BMI, is a measure of weight corrected for height (weight in kg/ [height in meters](to the second power)). Expected BMI is in the range of 22 to 24. Morbid obesity is defined as BMI greater than 44, and a BMI under 18 may be associated with anorexia. Other physical findings that in the opinion of the investigator would jeopardize the safety of the subject or the evaluation of the study objectives. A psychiatric condition, including schizophrenia, personality, anxiety, or affective disorders, which in the opinion of the investigator could compromise the subject's ability to participate in the trial. Known hypersensitivity to a component of the vaccine. Current drug or alcohol dependence as evidenced by a four-question screening interview to determine whether the subject has had medical, occupational, or family problems related to alcohol or illicit drug use during the past 12 months. These questions are derived from the Drug Abuse Screening Test (DAST-10) developed by the Addiction Research Foundation and recommended by the National Institute for Drug abuse as a tool for family physicians who wish to routinely screen new patients for drug abuse (http://www.nida.nih.gov/Diagnosis-Treatment/Diagnosis5.html). History of receipt of anthrax vaccine or history of diagnosis of or exposure to any form of anthrax. Member of the Armed Forces who deployed during Desert Storm/Desert Shield or who has been stationed in Korea or Southwest Asia since 1990, given the possibility of previous receipt of the licensed anthrax vaccine. Positive urine pregnancy test within the 24 hours prior to vaccination. Positive blood test for HIV, hepatitus B surface antigen or hepatitus C antibody, or syphilis (defined as positive RPR and FTA). Failure to pass the written exam. Employment in an industry involved in contact with large ruminant animals, such as working in a slaughter house, handling of raw animal hides or raw wool, veterinary sciences involving ruminant animals, or others where exposure to B. anthracis may occur. Screening laboratory values that fall outside the normal range as delineated in Appendix 3. Receipt of an experimental vaccine or medication within the 30 days prior to receipt of the study vaccine. Receipt of a live, attenuated vaccine within the 60 days prior to receipt of the study vaccine. Receipt of a subunit or killed vaccine within the 14 days prior to receipt of the study vaccine. Receipt of a blood product, including immunoglobulin, in the 90 days prior to receipt of the study vaccine. Anything that, in the opinion of the investigator, will compromise the participation of the subject with respect to his/her rights or risks. Oral temperature > 37.7 C or other acute illness occurring prior to inoculation on the day of vaccination. (This will lead to postponement of enrollment, not exclusion from the trial).

Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2003-07; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States